CLINICAL TRIAL: NCT00525863
Title: Oxygen Therapy in Schizophrenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Yuly Bersudsky, Ben Gurion University of the Negev
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BMHC-4602
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Schizophrenia
Keywords: schizophrenia; oxygen therapy
MeSH Terms: conditions — Schizophrenia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: oxygen — Patients will be treated with oxygen for 1 month and then for 1 month with regular air with the same flow rate and procedure or randomly in the opposite order. We propose to enrich the inspired oxygen partial pressure from 21 kPA to ~40 kPa in a double blind cross-over design. Ninety percent oxygen or regular air will be supplied from oxygen concentrators, through standard plastic nasal prongs, at a flow rate of 5 liters/minute, for 7 hours/day, throughout the night.

SUMMARY:
Due to intense ATP-consuming processes in the brain, a high level of brain energy supply is required. A popular hypothesis regarding the pathogenesis and pathophysiology of schizophrenia postulates hypofunction of neuronal circuits in the prefrontal and limbic-temporal areas. An emerging body of data suggests that impaired energy metabolism due to mitochondrial dysfunction plays a role in the pathophysiology of schizophrenia.

Under normal conditions cellular metabolic rate, i.e. oxygen and glucose consumption, increases proportionally with any increase in neuronal activity. The impaired energy metabolism due to mitochondrial dysfunction and frontal lobe hypofunction might be improved by increasing O2 supply to the brain. Oxygen-enriched air inhalation has been shown to increase brain oxygen supply. Hyperoxia therapy is a useful tool in the treatment of neurological and neurotrauma deficits.

We therefore suggest a randomized double blind cross-over study of enriched inspired O2 partial pressure in schizophrenia.

It is surprising given the numerous findings on reduced energy metabolism in schizophrenia that simple treatment with inspired enriched oxygen has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* 2 years of illness
* PANSS more than 60

Exclusion Criteria:

* unstable or serious physical illness
* suicidality
* drug abuse
* BMI above 30
* taking anti-hypertension medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
PANSS | every two weeks

SECONDARY OUTCOMES:
Clinical Global Impressions | every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yuly Bersudsky, MD, PhD, Principal Investigator — Ben-Gurion University of the Negev
Locations (1):
- Beersheva Mental Health Center, Beersheva, Israel